CLINICAL TRIAL: NCT05051553
Title: A Phase 1, Open-label, Single-center, 2-part Crossover Study to Evaluate the Relative Bioavailability of Fedratinib When Administered as Contents of Capsules Dispersed in a Nutritional Supplement Orally or Via Nasogastric Tube, or Administered Orally as Divided Doses of Intact Capsules With a Nutritional Supplement in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Bioavailability of Fedratinib When Administered in Different Ways to Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CA054-013
Expanded Access: NCT03723148 (Available)
Record Dates: First submitted 2021-09-16; First posted 2021-09-21 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers; Phase 1; Fedratinib
MeSH Terms: interventions — fedratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Treatment 1A (Experimental)
  Interventions: Drug: Fedratinib
- Treatment 1B (Experimental)
  Interventions: Drug: Fedratinib
- Treatment 2A (Experimental)
  Interventions: Drug: Fedratinib
- Treatment 2B (Experimental)
  Interventions: Drug: Fedratinib
- Treatment 2C (Experimental)
  Interventions: Drug: Fedratinib

INTERVENTIONS:
Drug: Fedratinib — Specified dose on specified days

SUMMARY:
The purpose of this study is to evaluate the relative bioavailability of fedratinib in healthy adult participants.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit: www.BMSStudyConnect.com

Inclusion Criteria:

* Body Mass Index (BMI) of 18.0 to 33.0 kg/m^2, inclusive. BMI = weight (kg)/(height [m])^2
* Healthy based on medical history, physical examination, clinical laboratory test results, vital signs, and 12-lead electrocardiogram (ECG) at screening and check-in

Exclusion Criteria:

* Allergy to or hypersensitive to any of the drugs or nutritional supplement used in the study
* Prior history of Wernicke's Encephalopathy
* Thiamine deficiency
* Hypersensitivity to ondansetron
* Has any medical condition, medical history, or use of concomitant medication that is contraindicated in the applicable drug labeling
* Has history, deviated nasal septum, and/or obstructed airway, bleeding disorders, or other inabilities for insertion of nasogastric (NG) tube (Part 2 only)

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
Fedratinib Pharmacokinetics: Estimation of maximum observed plasma concentration (Cmax) | Up to 12 days
Fedratinib Pharmacokinetics: Estimation of area under the curve (AUC) calculated from time zero to t, where t is the timepoint of the last quantifiable concentration (AUC(0-T)) | Up to 12 days
Fedratinib Pharmacokinetics: Estimation of AUC calculated from time zero extrapolated to infinite time (AUC(INF)) | Up to 12 days

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 66 days
Incidence of serious adverse events (SAEs) | Up to 66 days
Number of participants with clinically significant changes in electrocardiogram parameters | Up to 66 days
Incidence of clinically significant changes in vital signs: Body temperature | Up to 66 days
Incidence of clinically significant changes in vital signs: Respiratory rate | Up to 66 days
Incidence of clinically significant changes in vital signs: Blood pressure | Up to 66 days
Incidence of clinically significant changes in vital signs: Heart rate | Up to 66 days
Incidence of clinically significant changes in clinical laboratory results: Hematology tests | Up to 66 days
Incidence of clinically significant changes in clinical laboratory results: Clinical Chemistry tests | Up to 66 days
Incidence of clinically significant changes in clinical laboratory results: Urinalysis tests | Up to 66 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Syneos Health Clinical Research Services, Llc, Miami, Florida, United States

REFERENCES:
- [Derived] Chen Y, Wyatt D, Attanasio M, Thomas M, Thomas M, He B, Nishii R, Liu L, Shan V, Xue Y, Carayannopoulos LN, Ogasawara K, Krishna G. Relative bioavailability of fedratinib through various alternative oral administration methods in healthy adults. Cancer Chemother Pharmacol. 2024 Apr;93(4):307-317. doi: 10.1007/s00280-023-04612-w. Epub 2023 Nov 13. PMID 37955741
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm